CLINICAL TRIAL: NCT06286839
Title: An Open-Label Parallel Phase I Study Evaluating Multiple Ascending Dose Pharmacokinetics and Acute Immunomodulatory Potential of a Novel Oral Cannabidiol (CBD) Formulation
Brief Title: Study of Cannabidiol (CBD) in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NextEvo Inc. (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFCRO-150
Record Dates: First submitted 2023-10-07; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Immune System and Related Disorders; Immune System Diseases
Keywords: CBD; Phase 1; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Immune System Diseases | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 30 mg twice per day (Experimental): The 30mg dose will be consumed in 2 capsules twice per day, for 3 days and an extra 18 capsules in case of loss of study product
  Interventions: Dietary Supplement: Cannabidiol (CBD)
- 120 mg twice per day (Experimental): 120mg dose will be consumed in 8 capsules twice per day for 3 days and an extra 12 capsules in case of loss of study product
  Interventions: Dietary Supplement: Cannabidiol (CBD)

INTERVENTIONS:
Dietary Supplement: Cannabidiol (CBD) — Cannabidiol (CBD), a non-psychoactive component of Cannabis sativa L.

SUMMARY:
This was a prospective, single-centre, open label, randomized, two-arm, parallel design study to evaluate the effect of four-weeks consumption of active study product on primary endpoint in healthy adults

DETAILED DESCRIPTION:
Cannabidiol (CBD), a non-psychoactive component of Cannabis sativa L., has been purported to have a variety of beneficial physiological effects including but not limited to, pain relief, anti-anxiety, anti-seizure, anti-depressant, anti-oxidant, and anti-inflammatory. Despite the enthusiasm of the CBD industry for these claims, the empirical evidence supporting favourable physiological responses is inconsistent. These discrepancies may in part be explained by differences in CBD bioavailability when administered orally that in turn may be influenced by non-standardized CBD formulation, and/or the body size and composition of the recipient.

The purpose of this study was to test the bioavailability of two doses of a novel CBD formation given twice per day for three consecutive days in healthy study subjects and explore their potential acute anti-inflammatory properties as assessed by highly sensitive immunologic assays. The rationale for conducting the study was to evaluate the pharmacokinetic (PK) profile of a novel formulation of CBD designed to improve bioavailability given at two dose levels twice per day for three consecutive days. Although previous studies conducted in healthy study subjects have documented the safety and PK profile for a single dose of the test product, multiple ascending dose studies have not yet been conducted. In addition to evaluating multiple ascending dose PK, the pharmacodynamic properties of the CBD were assessed using ex vivo lipopolysaccharides (LPS) stimulated whole blood assays and high sensitivity serum cytokine assays.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent.
2. Be between 18 and 45, inclusive.
3. Has a BMI between 18-29.50 kg/m2.
4. Is in general good health, as determined by the investigator.
5. Willing to abstain from consuming tobacco or nicotine- containing products, consuming alcohol, grapefruit, or grapefruit juice, or taking any prescription drugs, dietary supplements, or non-prescription drugs for the periods required by the study protocol.
6. Willing to consume the investigational product daily for the duration of the trial.
7. Willing and able to communicate effectively with the study personnel and willing to comply with all protocol requirements, including visit schedule and oral intake of investigational product
8. Willing to consume the standard meal and an 8oz Boost nutritional drink at visit 2

Exclusion Criteria:

1. Are less than 18 or greater than 45
2. Participants who are pregnant or wish to become pregnant during the trial.
3. Participants who are lactating and/or currently breastfeeding
4. Post-menopausal, defined as one year without menses.
5. Participants currently of childbearing potential but not using an effective method of contraception, as outlined below:

   1. Complete abstinence from intercourse two weeks before administration of the investigational product, throughout the clinical trial, until the completion of follow-up procedures, or for two weeks following discontinuation of the investigational product in cases where the participant discontinues the trial prematurely. (Participants utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit).
   2. Has a male sexual partner who is surgically sterilized before the Screening Visit and is the only male sexual partner for that participant.
   3. Sexual partner(s) is/are exclusively female.
   4. Use of an acceptable method of contraception, such as a spermicide, mechanical barrier (e.g., male condom, female diaphragm), or contraceptive pill.

      The participant must use this method for at least 1 week before and 1 week following the end of the trial.
   5. Use of any intrauterine device (IUD) or contraceptive implant. The participant must have the device inserted at least 2 weeks before the first Screening Visit, throughout the trial, and 2 weeks following the end of the trial.
6. Are hypersensitive to any of the components of the investigational product.
7. Has taken any dietary supplement or non-prescription drugs within 3 days prior to baseline or has taken any prescription drugs within 14 days prior to baseline (antihistamines, acetaminophen, contraception or single- use over-the-counter medications including nonsteroidal anti-inflammatory drugs (NSAIDs) allowed before baseline.
8. Has a self-reported history of drug and/or alcohol abuse at the time of within 6 months before screening or exhibits evidence of drug and/or alcohol abuse at baseline.
9. Has consumed alcohol within 24 hours before screening and baseline.
10. Has consumed grapefruit or grapefruit juice within 3 days before screening or baseline
11. The participant has a current acute or chronic disease, which may, in the opinion of the investigator, impact the outcomes of the study.
12. The participant has clinically significant abnormal findings outside the normal screening ranges.
13. The participant has clinically significant abnormal findings from physical examination at screening and baseline that may, in the investigator's opinion, impact the study's outcomes.
14. The participant has a clinically important history of a medical disorder that may, in the opinion of the investigator, compromise the participant's safety or data quality
15. Current regular tobacco vape or nicotine-containing product use within 60 days prior to screening and between screening and baseline (Occasional use defined as less than 5 cigarettes per week or equivalent nicotine product/vape use)
16. Use of tetrahydrocannabinol (THC)/cannabidiol (CBD) products in within 7 days of screening.
17. The participant has a history of anaphylaxis, a documented hypersensitivity reaction, or a clinically important reaction to any drug which, in the opinion of the investigator, impacts the outcomes of the study.
18. A history of human immunodeficiency virus infection/acquired immune deficiency syndrome or a positive screening assessment for human immunodeficiency virus or viral hepatitis.
19. Evidence of amphetamines, barbiturates, Benzodiazepine (including prescription), cannabinoids, cocaine, opiates, phencyclidine, or ethanol on a urine drug screening at screening.
20. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
21. Participants may not be receiving treatment involving experimental drugs or devices. If the participant has been in a recent experimental trial, these must have been completed at least 30 prior to this trial.
22. Any Participant who is an employee of the investigational site an Atlantia Clinical Trials employee or their close family member, or a member of their household

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Plasma CBD pharmacokinetics of twice daily intake of 2 different doses of CBD over three days | T-30 minutes, T 0 minutes, T30 minutes, T60 minutes, T240 minutes (4 Hours), T480 minutes (8 Hours), and T4320 minutes (72 Hours)
  Difference in plasma CBD concentration (ng/ml) between groups as measured by total Area Under the Curve (tAUC) derived from plasma
Evaluate the safety of twice daily intake of 2 different doses of CBD over three 3 days | T-30 minutes, T 0 minutes, T30 minutes, T60 minutes, T240 minutes (4 Hours), T480 minutes (8 Hours), and T4320 minutes (72 Hours)
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Plasma CBD maximal concentration (Cmax, ng/ml) | T-30 minutes, T 0 minutes, T30 minutes, T60 minutes, T240 minutes (4 Hours), T480 minutes (8 Hours), and T4320 minutes (72 Hours)
  Difference in plasma Cmax concentration between groups as measured by total Area Under the Curve (tAUC) derived from plasma
Plasma CBD time to peak (Tmax, minutes) | T-30 minutes, T 0 minutes, T30 minutes, T60 minutes, T240 minutes (4 Hours), T480 minutes (8 Hours), and T4320 minutes (72 Hours)
  Difference in plasma Tmax concentration between groups as measured by total Area Under the Curve (tAUC) derived from plasma
Percentage Change between groups on whole blood LPS stimulated cytokines (% change) | T0 minutes, T4320 minutes(72 Hours)
  Differences between groups for the change from baseline were assessed for whole blood LPS stimulated cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Alice Eggleston, Principal Investigator — Atlantia Clinical Trials; David Chernoff, MD, Study Director — NextEvo Inc.
Locations (1):
- Altantia Clinical Trials, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
The data in this study will be published by NextEvo

REFERENCES:
- [Background] Millar SA, Stone NL, Yates AS, O'Sullivan SE. A Systematic Review on the Pharmacokinetics of Cannabidiol in Humans. Front Pharmacol. 2018 Nov 26;9:1365. doi: 10.3389/fphar.2018.01365. eCollection 2018. PMID 30534073
- [Background] Brunet LR, LaBrie S, Hagemann T. Immune monitoring technology primer: immunoprofiling of antigen-stimulated blood. J Immunother Cancer. 2016 Mar 15;4:18. doi: 10.1186/s40425-016-0122-4. eCollection 2016. No abstract available. PMID 26981248
- [Background] Hobbs JM, Vazquez AR, Remijan ND, Trotter RE, McMillan TV, Freedman KE, Wei Y, Woelfel KA, Arnold OR, Wolfe LM, Johnson SA, Weir TL. Evaluation of pharmacokinetics and acute anti-inflammatory potential of two oral cannabidiol preparations in healthy adults. Phytother Res. 2020 Jul;34(7):1696-1703. doi: 10.1002/ptr.6651. Epub 2020 Mar 8. PMID 32147925
- [Background] Williams NNB, Ewell TR, Abbotts KSS, Harms KJ, Woelfel KA, Dooley GP, Weir TL, Bell C. Comparison of Five Oral Cannabidiol Preparations in Adult Humans: Pharmacokinetics, Body Composition, and Heart Rate Variability. Pharmaceuticals (Basel). 2021 Jan 6;14(1):35. doi: 10.3390/ph14010035. PMID 33418866